CLINICAL TRIAL: NCT01924325
Title: Apixaban Versus Dual-antiplatelet Therapy (Clopidogrel and Aspirin) in High-risk Patients With Acute Non-disabling Cerebrovascular Events (ADANCE): Rationale, Objectives, and Design
Brief Title: Apixaban Versus Dual-antiplatelet Therapy (Clopidogrel and Aspirin) in Acute Non-disabling Cerebrovascular Events
Acronym: ADANCE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Xijing-ADANCE
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Ischemic Stroke; TIA
Keywords: apixaban; clopidogrel; aspirin; new oral anticoagulant; TIA; acute minor ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — apixaban; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dual-antiplatelet Therapy (Active Comparator): Receiving a 75 mg dose of clopidogrel and 75mg dose of aspirin from day 1 to day 21, with placebo apixaban twice daily
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Drug: placebo
- Apixaban 2.5mg (Experimental): Receiving a 2.5-mg twice daily of apixaban, with placebo clopidogrel and placebo aspirin from day 1 to day 21
  Interventions: Drug: Apixaban; Drug: placebo
- Apixaban 5mg (Experimental): Receiving a 5-mg twice daily of apixaban, with placebo clopidogrel and placebo aspirin from day 1 to day 21
  Interventions: Drug: Apixaban; Drug: placebo

INTERVENTIONS:
Drug: Apixaban — orally active direct factor Xa inhibitor
  Other Names: Eliquis; BMS-562247; BMS-562247-01
  Arms: Apixaban 2.5mg; Apixaban 5mg
Drug: Clopidogrel — an irreversible inhibitor of the P2Y12 adenosine diphosphate receptor
  Other Names: Plavix; Clopivid
  Arms: Dual-antiplatelet Therapy
Drug: Aspirin — a non-steroidal anti-inflammatory drug
  Other Names: Acetylsalicylic acid
  Arms: Dual-antiplatelet Therapy
Drug: placebo

SUMMARY:
Nondisabling cerebrovascular events represent the largest group of cerebrovascular disease with a high risk of recurrent stroke. A recent trial indicated that clopidogrel and aspirin treatment reduced the risk of recurrent stroke and was not associated with increased hemorrhage events, compared with aspirin monotherapy. Apixaban, a new oral anticoagulant, is proved to be as effective as traditional anticoagulants with less risk of bleeding events.

To estimate whether apixaban is beneficial for acute TIA or minor stroke, a randomized, double-blind, multicenter, controlled clinical trial has been designed. The investigators will assess the hypothesis that a 21-days apixaban regimen is superior to clopidogrel and aspirin dual-therapy for the treatment of high-risk patients with acute nondisabling cerebrovascular event.

DETAILED DESCRIPTION:
The ADANCE study is a randomized, double-blind clinical trial with a target enrollment of 3,000 Chinese patients. Two subtypes of patients will be enrolled: I, acute disabling ischemic stroke (<24 hours of symptoms onset); II, acute TIA (<24 hours of symptoms onset).

Patients will be randomized into 3 groups:

Ⅰ Receiving a 75 mg dose of clopidogrel and 75mg dose of aspirin from day 1 to day 21, with placebo apixaban twice daily.

Ⅱ Receiving a 2.5-mg twice daily of apixaban, with placebo clopidogrel and placebo aspirin from day 1 to day 21.

Ⅲ Receiving a 5-mg twice daily of apixaban, with placebo clopidogrel and placebo aspirin from day 1 to day 21.

From day 22 to 3 months, all patients will receive 75-mg dose of clopidogrel long-term antiplatelet therapy.

The primary efficacy end point is percentage of patients with new stroke (ischemic or hemorrhage) at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (male or female ≥18 years old)
* Acute nondisabling ischemic stroke (NIHSS ≤3 at the time of randomization) that can be treated with study drug within 24 hours of symptoms onset. Symptom onset is defined by the "last see normal" principle
* TIA (neurologic deficit attributed to focal brain ischemia, with resolution of the deficit within 24 hours of symptom onset), that can be treated with investigational medication within 24 hours of symptoms onset. Symptom onset is defined by the "last see normal" principle
* Informed consent signed

Exclusion Criteria:

* Diagnosis of hemorrhage or other pathology, such as vascular malformation, tumor, abscess or other major nonischemic brain disease, on baseline head CT or MRI scan
* mRS score >2 at randomization (premorbid historical assessment) NIHSS ≥4 at randomization
* Clear indication for anticoagulation (atrial fibrillation, mechanical cardiac valves, deep venous thrombosis, pulmonary embolism or known hypercoagulable state)
* Contraindication to investigational medications
* Thrombolysis for ischemic stroke within preceding 7 days
* History of intracranial hemorrhage
* Current treatment (last dose given within 10 days before randomization) with heparin therapy or oral anticoagulation
* Gastrointestinal bleed or major surgery within 3 months
* Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months
* TIA or minor stroke induced by angiography or surgery
* Severe noncardiovascular comorbidity with life expectancy <3 months
* Women of childbearing age not practicing reliable contraception who do not have a documented negative pregnancy test result
* Severe renal failure, defined as Glomerular Filtration Rate (GFR) <30 ml/min Severe hepatic insufficiency (Child-Pugh score B to C)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with new stroke (ischemic or hemorrhage) | 90 days

SECONDARY OUTCOMES:
Percentage of patients with new clinical vascular events (ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/vascular death) | 30 days
Percentage of patients with new clinical vascular events (ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/vascular death) | 30 days and 90 days
Changes in NIHSS scores | 90 days
moderate to severe bleeding events | 90 days
Total mortality | 90 days
Adverse events/severe adverse events reported by the investigators | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, M.D., Principal Investigator — Neurology Department,Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China